CLINICAL TRIAL: NCT01638871
Title: Internet-Based Osteoarthritis Pain Coping Skills Intervention
Acronym: PainCOACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-1384; 5R01AR057346-02 (NIH)
Record Dates: First submitted 2012-06-21; First posted 2012-07-12 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2014-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Study arm will complete the 8-week Internet-based pain coping skills program.
  Interventions: Behavioral: PainCOACH
- Control Group (No Intervention): This study arm will only provide demographic and pain-related information.

INTERVENTIONS:
Behavioral: PainCOACH — The 8-week Internet-based pain coping skills intervention program includes 8 sessions. Each session takes 30-45 minutes to complete and includes text, illustrations, photos, animations, audio narration, interactivity, and delivery of personalized feedback. Users will be expected to complete 1 session per week.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to translate a proven pain coping skills intervention for osteoarthritis (OA) patients into an engaging and easy-to-use Internet-based intervention that uses innovative technologies to mimic traditional, in-person training sessions.

DETAILED DESCRIPTION:
Twenty-one million Americans live with osteoarthritis (OA), a progressive joint disease that causes stiffness, pain, reduced range of motion, distress, and decrements in physical, social, and role functioning. Medical treatments for OA pain are limited and present risks, especially for older populations. However, cognitive behavioral pain coping skills interventions have proven effective for decreasing OA pain, disability, and distress. Unfortunately, existing programs reach a limited number of patients because they require patients to travel to receive in-person training. There is a need for interventions that address the needs of a larger proportion of the rapidly growing population of people whose functioning and quality of life are severely diminished by OA. Delivering proven pain management interventions via the Internet is a promising way to address this need, especially in light of increasing use of the Internet by older Americans. To be most effective, an Internet-based intervention would need to mimic key features of in-person interventions. The proposed intervention will do that by translating a proven in-person pain coping skills protocol into an interactive Internet-based application that uses multimedia and expert systems technology to mimic in-person interventions. It will provide individualized feedback, interactive problem solving, and animated demonstrations, and it will incorporate learning techniques from Bandura's Social Cognitive Theory, including modeling, mastery experiences, and social reinforcement. The project includes two phases, corresponding to two specific aims. In Phase I the investigators will translate the in-person intervention for delivery on the Internet. This phase will including gathering feedback from patient and expert therapist focus groups, which will help refine the program. In Phase II the investigators will conduct a small-scale randomized controlled trial that will enable us to examine and refine features designed to increase motivation and adherence over the course of the 8-week Internet-based intervention. The trial will also enable the investigators to demonstrate its feasibility, tolerability, safety, and promise. The investigators hypothesize that the trial will demonstrate the effectiveness of the Internet for delivery of this OA pain coping skills intervention. Taken together, these activities will prepare the program for testing in a full-scale randomized controlled trial in the next stage of this research. The promise of this project is enhanced by the multi-disciplinary research team, which has expertise in the conduct of cognitive behavioral interventions that teach OA patients to use coping skills to manage their pain, developing and implementing individualized computerized feedback reports using expert systems technology, and development of engaging, user-friendly, interactive computer-based programs for learning and assessment. Relevance: This Internet-based OA pain coping skills intervention targets a significant individual and public health problem and expands access to an empirically-supported pain self-management program so that it can reach a greater proportion of the large and growing population of people suffering from OA pain and related disability.

ELIGIBILITY:
Inclusion Criteria:

* A formal clinical diagnosis of OA affecting one or both knees or hips
* Significant OA pain
* Must be aged 18 or older
* Must be English speaking

Exclusion Criteria:

* Not fluent in English
* Have less than 7th grade English reading proficiency
* Show signs of cognitive impairment that would prevent comprehension of consent procedures or study measures and procedures
* Have a medical condition that would contraindicate safe participation in the study (as determined by study physician)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity | Baseline to post-intervention (at approximately 10 weeks and at 6 months)
  The Arthritis Impact Measurement Scale-2 (AIMS-2) pain subscale that measures severity of arthritis pain, frequency of severe pain, duration of morning stiffness, frequency of joint pain, and difficulty sleeping due to pain

SECONDARY OUTCOMES:
Change in pain-related anxiety | Baseline to post-intervention (at approximately 10 weeks and at 6 months)
  Pain Anxiety Symptoms Scale, 20 item version (PASS-20), which assesses fear of pain, cognitive anxiety, escape-avoidance behaviors, and physiological symptoms of anxiety
Change in pain-related interference with functioning | Baseline to post-intervention (at approximately 10 weeks and at 6 months)
  Arthritis Impact Measurement Scale-2 (AIMS-2) functioning subscales, summed across mobility, walking/bending, self- care, household tasks, social activities, work activities
Change in bodily relaxation | Baseline to post-intervention (at approximately 10 weeks)
  From a behavioral observation task; assessed with brief self-report measure of perceived relaxation and electromyograph (EMG) monitor using external electrodes measuring frontalis muscle tension and indicated by change in frontalis muscle tension during the relaxation task and muscle tension achieved at end of task
Change in problem solving skills | Baseline to post-intervention (at approximately 10 weeks)
  From a behavioral observation task; quality and quantity of responses to hypothetical situation describing a pain flare and asking participants how they would manage it, along with subjective success assessed with an adapted version of the Arthritis Self-Efficacy scale (ASE)
Change in emotional adjustment | Baseline to post-intervention (at approximately 10 weeks)
  Positive and Negative Affect Schedule-20 item version (PANAS)
Program Usability | Post-intervention (at approximately 10 weeks)
  To help assess tolerability of the intervention site; for intervention arm participants only; qualitative (open-ended) questions to gather feedback on PainCOACH program (usability, usefulness, influence on attitudes/motivation, likes/dislikes)
Number of participants recruited | up to 10 weeks
  To assess feasibility
Number of participants who complete the study | through 10 weeks and/or 6 months
  To assess tolerability
Number of participants who adhere to study protocol | through 10 weeks and/or 6 months
  To assess tolerability
Medication type and frequency of use during the past week | Baseline, mid-point, and post-intervention
  To help assess types of medication used for arthritis pain
Change in and use of pain coping strategies | Baseline to post-intervention (at approximately 10 weeks and at 6 months)
  Adapted Coping Strategies Questionnaire (CSQ), Chronic Pain Coping Inventory (CPCI) subscales, West Haven-Yale Multidimensional Pain Inventory (WHYMPI) subscales, and additional items that measure use of strategies taught
Personality | Baseline
  Ten-Item Personality Inventory (TIPI)
Change in self-efficacy for pain management | Baseline to post-intervention (at approximately 10 weeks and at 6 months)
  Arthritis Self-Efficacy scale (ASE)
Change in social support | Baseline to post-intervention (at approximately 10 weeks)
  Adapted West Haven-Yale Multidimensional Pain Inventory (WHYMPI) subscale

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rini, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - UNC-CH Thurston Arthritis Research Center, Smithfield, North Carolina